CLINICAL TRIAL: NCT04092387
Title: Low Nicotine Content Cigarettes in Vulnerable Populations: Women of Reproductive Age
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Food and Drug Administration (FDA) (U.S. Federal Agency); Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Stephen T. Higgins, PhD, Professor, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CHRMS19-0129; U54DA036114-06 (NIH)
Record Dates: First submitted 2019-09-13; First posted 2019-09-17 (Actual); Results first posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Tobacco Use Disorder
Keywords: Biomarkers of Exposure; Nicotine Dependence; Reduced Nicotine Cigarettes; Tobacco Withdrawal; Women; Health Disparities; Vulnerable Populations; E-Cigarettes
MeSH Terms: conditions — Tobacco Use Disorder; Vaping | interventions — Electronic Nicotine Delivery Systems

STUDY DESIGN:
Intervention Model Description: Randomized parallel groups research design.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double blind dosing of tobacco cigarette nicotine content levels.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- RC 1 only (Experimental): Research cigarettes #1
  Interventions: Other: Varying the nicotine content of cigarettes
- RC 2 only (Experimental): Research Cigarettes #2
  Interventions: Other: Varying the nicotine content of cigarettes
- RC 2 + EC 1 (Experimental): Research Cigarettes #2 plus E-cigarettes #1
  Interventions: Other: Varying the nicotine content of cigarettes; Other: E-Cigarettes
- RC 2 + EC 2 (Experimental): Research Cigarettes #2 plus E-cigarettes #2
  Interventions: Other: Varying the nicotine content of cigarettes; Other: E-Cigarettes

INTERVENTIONS:
Other: Varying the nicotine content of cigarettes — 1) Altering the nicotine content of the tobacco research cigarettes
  Other Names: Comparing normal nicotine content (RC1) to very low nicotine content (RC2)
Other: E-Cigarettes — Comparing effects of combining RC2 with EC 1 versus EC2
  Other Names: e-cigarette with only tobacco flavor (EC 1); e-cigarette in multiple flavors ( EC2)
  Arms: RC 2 + EC 1; RC 2 + EC 2

SUMMARY:
Despite marked reductions in cigarette smoking in the general population, smoking among economically disadvantaged women has increased. Smoking among women of reproductive age is a particular concern because in addition to the usual health risks, there are additional risks should they become pregnant. A national nicotine reduction policy for cigarettes has considerable potential to reduce tobacco use, dependence, and improve health in this population. Controlled trials in general population samples have demonstrated that reducing the nicotine content in cigarettes can reduce cigarettes per day (CPD), dependence severity, and tobacco toxicant exposure.

The goal of the proposed trial is to experimentally examine whether increasing the availability and appeal of an alternative, non-combusted source of nicotine (e-cigarettes) enhances the effect of altering the nicotine in cigarettes in non-pregnant female cigarette smokers of childbearing age. Additionally, investigators will test whether allowing participants to personalize the flavor of the e-liquid alters any moderating effects their availability may have on tobacco cigarette smoking.

Daily smokers who are female, aged 21-44 years, and have a maximum educational attainment of graduating high school, will be recruited at Johns Hopkins University and the University of Vermont.

Investigators will study two research cigarettes referred to here as Research Cigarettes 1 (RC1) and Research Cigarettes 2 (RC2). One will be a normal nicotine content cigarette and the other a reduced nicotine content cigarette. Investigators will study two e-cigarette conditions referred to here as E-Cigarette Condition 1 (EC1) and E-Cigarette Condition 2 (EC2). Both e-cigarette conditions will involve the same commercially available devices and same nicotine-containing e-liquid, but in one condition that e-liquid will be available only in tobacco flavor while in the other the e-liquid will be available in multiple flavors from which participants can choose three based on personal preference. Participants will be assigned to one of the following four conditions: (1) RC1 only; (2) RC2 only; (3) RC2 + EC1; (4) RC2 + EC2.

Participants will be asked to use only their assigned study products for 16 weeks. Outcome measures include total CPD, craving, withdrawal, psychiatric symptoms, breath carbon monoxide (CO), other biomarkers of tobacco toxicant exposure, and cigarette demand assessed by behavioral economic purchase tasks.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 21 to 44 years old

Exclusion Criteria:

* Male
* Under 21 years old
* Over 44 years old

Ages: 21 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participants must be female.
Enrollment: 326 (Actual)
Dates: Start 2020-10-18 (Actual); Primary Completion 2023-11-27 (Actual); Study Completion 2023-11-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen T. Higgins, Ph.D., Principal Investigator — University of Vermont
Locations (2):
- United States (2):
  - Johns Hopkins University, Baltimore, Maryland
  - University of Vermont, Burlington, Vermont

IPD SHARING:
Plan to Share IPD: Yes
de-identified data
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available once we have published the results of the parent trials and manuscripts based on secondary analyses of those data, which we anticipate taking approximately three years
Access Criteria: request data for stated scientific purpose

REFERENCES:
- [Derived] Higgins ST, Sigmon SC, Tidey JW, Heil SH, Gaalema DE, Lee DC, DeSarno MJ, Klemperer EM, Menson KE, Cioe PA, Plucinski S, Wiley RC, Orr E. Reduced Nicotine Cigarettes and E-Cigarettes in High-Risk Populations: 3 Randomized Clinical Trials. JAMA Netw Open. 2024 Sep 3;7(9):e2431731. doi: 10.1001/jamanetworkopen.2024.31731. PMID 39240566

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RC 1 Only | RC 2 Only | RC 2 + EC 1 | RC 2 + EC 2
Started | 83 | 85 | 74 | 84
Completed | 67 | 66 | 57 | 70
Not Completed | 16 | 19 | 17 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RC 1 Only | RC 2 Only | RC 2 + EC 1 | RC 2 + EC 2 | Total
Number analyzed (Participants) | 83 | 85 | 74 | 84 | 326
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.77 (10.98) | 39.85 (9.28) | 41.51 (12.39) | 39.38 (10.59) | 40.09 (10.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 69 | 50 | 59 | 243
  Male | 18 | 16 | 24 | 25 | 83
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black, non-Latino | 9 | 6 | 9 | 9 | 33
  Latino | 4 | 3 | 3 | 2 | 12
  White, non-Latino | 66 | 68 | 60 | 68 | 262
  Non-Latino other or multiracial | 4 | 8 | 2 | 5 | 19
Region of Enrollment [Number; unit: participants]
  United States | 83 | 85 | 74 | 84 | 326
Population [Count of Participants; unit: Participants]
  Females with lower educational level | 20 | 23 | 16 | 21 | 80
  OUD | 19 | 19 | 17 | 19 | 74
  Affective disorders | 44 | 43 | 41 | 44 | 172
Educational level [Count of Participants; unit: Participants]
  <High school | 9 | 4 | 3 | 14 | 30
  High school graduate, equivalency, or some college | 51 | 57 | 46 | 47 | 201
  Associate's degree | 8 | 11 | 13 | 11 | 43
  ≥College graduate | 15 | 13 | 12 | 12 | 52
Marital status [Count of Participants; unit: Participants]
  Married | 8 | 15 | 17 | 11 | 51
  Never married | 49 | 47 | 36 | 48 | 180
  Divorced, separated, or widowed | 26 | 23 | 21 | 25 | 95
Primarily smokes mentholated cigarettes [Count of Participants; unit: Participants] | 32 | 35 | 31 | 33 | 131
Cigarettes smoked per day [Mean (Standard Deviation); unit: cigarettes per day] | 16.42 (8.02) | 18.44 (9.47) | 17.86 (9.11) | 16.90 (8.85) | 17.40 (8.87)
Urine cotinine level [Mean (Standard Deviation); unit: ng/mL] | 4499.25 (3120.20) | 5235.67 (3251.28) | 5156.57 (4150.44) | 5293.33 (3799.45) | 5043.55 (3680.12)
Breath CO level [Mean (Standard Deviation); unit: ppm] | 20.90 (14.02) | 19.30 (12.39) | 21.03 (13.38) | 20.66 (13.44) | 20.46 (13.28)
Age started smoking regularly [Mean (Standard Deviation); unit: years] | 16.61 (3.97) | 15.92 (3.91) | 16.24 (3.84) | 16.79 (5.15) | 16.39 (4.26)
FTND score [Mean (Standard Deviation); unit: scores on a scale] — Fagerstrom Test for Nicotine Dependence:
  In scoring the Fagerstrom Test for Nicotine Dependence, the three yes/no items are scored 0 (no) and 1 (yes). The three multiple-choice items are scored from 0 to 3.
  The items are summed to yield a total score of 0-10.
  Classification of dependence, based on total score:
  0-2 Very low 3-4 Low 5 Moderate 6-7 High 8-10 Very high
  scores on a scale | 5.12 (2.24) | 5.31 (2.20) | 5.26 (2.31) | 4.70 (2.07) | 5.09 (2.21)
Used other tobacco products, past 30 days [Count of Participants; unit: Participants] | 5 | 4 | 5 | 9 | 23
Used e-cigarettes, past 30 days [Count of Participants; unit: Participants] | 13 | 11 | 5 | 13 | 42

OUTCOME MEASURES:

1. Primary Outcome: Number of Cigarettes Smoked Per Day
Description: Cigarettes per day will be assessed for use of cigarettes with different nicotine content.
Time Frame: 16 weeks
Population: Participants who completed week 16 of study
Measure: Least Squares Mean (Standard Error); unit: cigarettes per day
Arm/Group | RC 1 Only | RC 2 Only | RC 2 + EC 1 | RC 2 + EC 2
Number analyzed (Participants) | 67 | 66 | 57 | 70
cigarettes per day | 22.54 (1.59) | 14.32 (1.32) | 11.76 (1.18) | 7.63 (0.90)

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | RC 1 Only | RC 2 Only | RC 2 + EC 1 | RC 2 + EC 2
All-Cause Mortality (participants affected / at risk) | 0/83 | 0/85 | 1/74 | 0/84
Serious Adverse Events (participants affected / at risk) | 9/83 | 4/85 | 4/74 | 2/84
Other Adverse Events (participants affected / at risk) | 71/83 | 74/85 | 62/74 | 72/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RC 1 Only (N=83) | RC 2 Only (N=85) | RC 2 + EC 1 (N=74) | RC 2 + EC 2 (N=84)
Psychiatric disorders - Other (Psychiatric disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Esophageal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Irritability (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pregnancy, puerperium and perinatal conditions (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Surgical and medical procedures - Other (Surgical and medical procedures) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal calculi (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Death NOS (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RC 1 Only (N=83) | RC 2 Only (N=85) | RC 2 + EC 1 (N=74) | RC 2 + EC 2 (N=84)
OASIS Score Increase (Psychiatric disorders) | 32 (51) | 31 (43) | 31 (42) | 31 (40)
BDI Category Increase (Psychiatric disorders) | 29 (51) | 29 (40) | 26 (34) | 25 (41)
Psychiatric disorders (Psychiatric disorders) | 27 (53) | 28 (43) | 19 (27) | 24 (37)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 23 (38) | 27 (44) | 18 (40) | 18 (35)
General disorders and administration (General disorders) | 18 (25) | 24 (27) | 16 (20) | 22 (27)
Infections and infestations (Infections and infestations) | 16 (17) | 23 (24) | 8 (11) | 10 (13)
Nervous system disorders (Nervous system disorders) | 7 (8) | 18 (23) | 15 (19) | 10 (11)
Gastrointestinal disorders (Gastrointestinal disorders) | 9 (14) | 17 (25) | 14 (20) | 17 (23)
Vascular disorders (Vascular disorders) | 10 (13) | 13 (15) | 8 (10) | 16 (30)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 11 (14) | 16 (16) | 7 (7) | 12 (12)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 6 (7) | 4 (7) | 4 (4) | 5 (8)
Surgical and medical procedures (Surgical and medical procedures) | 2 (2) | 3 (3) | 5 (5) | 4 (4)
Cardiac disorders (Cardiac disorders) | 4 (6) | 2 (4) | 3 (4) | 3 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-01-23): https://cdn.clinicaltrials.gov/large-docs/87/NCT04092387/Prot_SAP_000.pdf
  • Informed Consent Form (2023-01-23): https://cdn.clinicaltrials.gov/large-docs/87/NCT04092387/ICF_001.pdf